CLINICAL TRIAL: NCT06098404
Title: Correlates of CRCI and Gut Microbiome Dysbiosis; a Pilot Study
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0289
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Microbiome; Fatigue; Cognition
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood and Stool will be coll
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer Patients: Patients diagnosed with cancer undergoing standard of care treatment.

SUMMARY:
The aim of this study is to characterize the microbiome and assess fatigue and cognition of patients with cancer undergoing standard of care treatment.

DETAILED DESCRIPTION:
Cancer-related fatigue is experienced by nearly all patients during treatment, and cancer-related cognitive impairment (CRCI), which is a decrease in neurocognitive functioning that can be caused by cancer or its treatment, is present in up to ¾ of patients during treatment. Fatigue and CRCI have both been linked to the composition of the gut microbiome in cancer patients. CRCI is often reported as one of the most debilitating and life-altering aspects of cancer and treatment. Although CRCI is widely reported in patients with a variety of cancers and undergoing a variety of treatments, it is not clear if the mechanisms leading to symptoms are the same throughout. Using identical methods to monitor CRCI symptoms and microbial dysbiosis in a cross-section of various cancers, cancer stages, and treatments, can help to identify commonalities associated with symptoms.

Specific Aims

Specific Aim 1: Characterize the microbiome of cancer patients and compare to healthy control subjects from previous studies.

Specific Aim 2: Assess fatigue in cancer patients and determine associations with composition of the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of cancer.
2. Ages 18 and over.
3. Has access to a device (smart phone, computer, tablet) with internet access.
4. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Other medical conditions or medications deemed exclusionary by the study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from community cancer clinics
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Characterization of fecal microbiome using molecular methods at baseline | Baseline
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for PCR at baseline
Characterization of fecal microbiome using molecular methods at 6 months | 6 months
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for PCR after 6 months of standard of care treatment.

SECONDARY OUTCOMES:
Cognitive Function as measured by Montreal Cognitive Assessment at baseline | Baseline
  The Montreal Cognitive Assessment (MoCA) is a rapid assessment of cognition. The MoCA-BLIND v8.1 will be used in this study as it can be administered in person as well as over the telephone. The MoCA-BLIND consists of 9 questions with the following subcategories: memory, attention, language, abstraction, delayed recall and orientation. The MoCA has been used extensively to detect cognitive impairment in many conditions, including head trauma. The MoCA will be administered by a certified tester at enrollment. Scores range from 0 to 22, higher score being a better outcome.
Cognitive Function as measured by Montreal Cognitive Assessment at 6 months | 6 months
  The Montreal Cognitive Assessment (MoCA) is a rapid assessment of cognition. The MoCA-BLIND v8.2 will be used in this study as it can be administered in person as well as over the telephone. The MoCA-BLIND consists of 9 questions with the following subcategories: memory, attention, language, abstraction, delayed recall and orientation. The MoCA has been used extensively to detect cognitive impairment in many conditions, including head trauma. The MoCA will be administered by a certified tester at enrollment. Scores range from 0 to 22, higher score being a better outcome. The MoCA will be performed after 6 months of standard of care treatment.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale at baseline | Baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale at 6 months | 6 months
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition. The FACS will be performed after 6 months of standard of care treatment.
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at baseline | Baseline
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at 6 months. | 6 months
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome). The GSRS will be performed after 6 months of standard of care treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No